CLINICAL TRIAL: NCT05463315
Title: A Mixed Methods Sequential Explanatory Study to Evaluate the Effectiveness of Applying Moziak Device Compared to Standard Manual Compression on Arterio-Venous Fistula Puncture Sites Haemostasis
Brief Title: Applying Moziak Device Compared to Standard Manual Compression on Arterio-Venous Fistula Puncture Sites Haemostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Magda Bayoumi, Assisstant Professor, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NURSING119
Record Dates: First submitted 2022-07-15; First posted 2022-07-18 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Post Dialysis Arterio-Venous Fistula Puncture Sites

STUDY DESIGN:
Intervention Model Description: A Mixed Methods Sequential Explanatory Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moziak Device (Experimental): Applying Moziak Device Compared to Standard Manual Compression
  Interventions: Device: Moziak Device

INTERVENTIONS:
Device: Moziak Device — Applying Moziak Device Compared to Standard Manual Compression
  Other Names: Standard Manual Compression

SUMMARY:
The study aimed to evaluate the Effectiveness of Applying Moziak Device Compared to Standard Manual Compression Post Dialysis Arterio-Venous Fistula Puncture Sites Haemostasis

DETAILED DESCRIPTION:
application of new device to find a Solution for Nursing Challenge for caring patient Post Dialysis Arterio-Venous Fistula Puncture Sites Haemostasis

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing hemodialysis therapy
* Both sex

Exclusion Criteria:

* Less than 18 years old
* Patient has central vascular access

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change the time of Haemostasis post dialysis | 3 months
  Applying Moziak Device Compared to Standard Manual Compression Post Dialysis Arterio-Venous Fistula Puncture Sites

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No